CLINICAL TRIAL: NCT01467817
Title: Obesity/Overweight in Persons With Early and Chronic SCI: A Randomized Multi-Center Controlled Lifestyle Intervention
Brief Title: Obesity/Overweight in Persons With Early and Chronic Spinal Cord Injury (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TMP-MN-009
Record Dates: First submitted 2011-09-26; First posted 2011-11-09 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-02

CONDITIONS: Overweight; Obese; Spinal Cord Injury
Keywords: body mass; abdominal fat; whole body lean mass; insulin resistance; caloric intake; expenditure; endurance; Strength; TC:HDL ratio; LDL:HDL ratio; area under the TG response curve; feeding challenge; fasting and post-prandial whole body fat oxidation; HRQoL
MeSH Terms: conditions — Overweight; Obesity; Spinal Cord Injuries; Insulin Resistance; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Intervention (Experimental): This arm will test the combination of 6 months of structured lifestyle intervention incorporating education, exercise, diet, and behavioral support.
  Interventions: Behavioral: Lifestyle Intervention
- Exercise Control (Placebo Comparator): This arm will test the benefits of exercise alone while controlling for investigator contact.
  Interventions: Behavioral: Exercise Control

INTERVENTIONS:
Behavioral: Lifestyle Intervention — The intervention incorporates 6 months of active structured lifestyle intervention containing participant education, exercise, dietary intervention, and behavioral support
  Arms: Lifestyle Intervention
Behavioral: Exercise Control — The control group intervention will test benefits of exercise alone while controlling for investigator contact.
  Arms: Exercise Control

SUMMARY:
The purpose of this study is to determine how exercise and nutritional guidance and supplementation affects your physical fitness, risk for heart disease, your body's ability to burn fat, and your opinions about your health.

DETAILED DESCRIPTION:
The study plan will enroll 80 persons with Spinal Cord Injury (SCI) who are overweight/obese and have fasting atherogenic dyslipidemia and dysglycemia. A Data Safety Management Board will oversee the trial. Interventions will include 6 months of structured lifestyle intervention incorporating education, exercise, diet, and behavioral support A second arm will test benefits of exercise alone while controlling for investigator contact. Multiple baselines tested before intervention will serve as a treatment control.

Exercise will include a six-month circuit resistance training program already established as effective in fitness attainment for persons with paraplegia and tetraplegia. Dietary intervention over the same period will balance caloric expenditure measured by indirect calorimetry and food intake, the latter coming from a Mediterranean style diet having effectiveness established in the DPP for durable weight loss and diabetes prevention. The investigators and personal 'lifestyle coaches' will then shape and follow client-specific exercise and diet programs to be conducted for 12 months in the home or community-based centers. Behavioral approaches will include a 16-week training curriculum presented in both small groups and with the lifestyle coaches. Other behavioral approaches will include customized trial information booklets, performance incentives, outcome challenges between centers, and use of the VA Telehealth system for performance tracking, compliance assessment, and motivational support.

Study specific aims and their accompanying hypotheses will test effects of intervention on: 1) reducing body weight and radiographically-derived body fat, 2) improving fitness as assessed by endurance, strength, and anaerobic power, 3) reducing risks of fasting dyslipidemia, post-prandial lipemia, and insulin resistance, and 4) enhancing perceived health-related quality of life. Data will be analyzed by Multivariate analysis with repeated measures. Ancillary testing will investigate effects of intervention on the whole body oxidation of fat at rest and following food intake, and examine the relationship between dietary intake and caloric expenditure at the beginning and the end of the 18 month study. The primary trial goal pays fidelity to the DPP by targeting sustained loss of 7% of body weight, a proven countermeasure for prevention of diabetes. Positive results of training will represent the first evidence-based randomized multi-center trial of sustained weight loss in persons with SCI - military or civilian. In the near term the data will provide evidence needed to initiate health reform of military and non-military constituencies with disability. The information will also underwrite changes in dietary support of newly injured persons. The information will further provide a roadmap for clinicians to institute client-centered programs of health planning and recovery. As the extension phase will test both home and community-based programs, deployment to wider military constituencies of persons with SCI can be achieved through VA Community Outpatient Clinics. The trial can also become a roadmap to weight and disease management experience by persons with physical impairments other than SCI.

ELIGIBILITY:
Inclusion Criteria:

* participants will include 64 men and women aged 18-65 years with SCI (AIS A-C) at the C5-L1 levels for more than 1 year.
* the International Standards for Neurological Classification of SCI (ASIA/ISCoS) will serve as benchmarks for subject classification. A physician-rater experienced in these procedures will classify subjects upon study entry.

Exclusion Criteria:

Study candidates will be excluded from study because of:

* structured exercise conditioning for recreation or competition within 6 months of study entry;
* defined diet involving caloric restriction or nutrient modification;
* weight loss or gain of 5% within the preceding 6 months;
* surgery within 6 months;
* pressure ulcer within 3 months;
* upper limb pain that limits exercise;
* recurrent acute infection or illness requiring hospitalization or IV antibiotics;
* pregnancy;
* previous MI or cardiac surgery;
* 6 month history of glucose-lowering and lipid-lowering drug therapy;
* Type I or II diabetes (by WHO criteria); and
* daily intake of vitamin supplements exceeding 100% RDA.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Body mass | 12 months
  Study specific aims and their accompanying hypotheses will test effect of intervention on:1)reducing body weight and radiographically-derived body fat, 2)improving fitness as assessed by endurance, strength, and anaerobic power,3) reducing risks of fasting dyslipidemia, post-prandial lipemia, and insulin resistance, and 4) enhancing perceived health-related quality of life. the primary trial goal pays fidelity to the DPP by targeting sustained loss of 7% of body weight, a proven countermeasure for prevention of diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami
Locations (1):
- University Of Miami, Miami, Florida, United States

REFERENCES:
- See also: Related Info — http://www.themiamiproject.org